CLINICAL TRIAL: NCT06192511
Title: Implementing a Novel Consent Process for Biospecimen Research After Newborn Screening in Hospitals Serving Diverse Patients
Brief Title: Implementing a Novel Consent Process for Biospecimen Research After Newborn Screening
Acronym: MICI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erin Rothwell (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Erin Rothwell, Professor, University of Utah
Organization: University of Utah (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 00153608
Record Dates: First submitted 2023-12-04; First posted 2024-01-05 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Implementation Science; Informed Consent; Neonatal Screening
Keywords: newborn screening; informed consent; biobanking
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (No Intervention): Standard education provided about the Michigan BioTrust includes a brief verbal description from hospital staff and a brochure. Materials will be provided in English, Spanish, or Arabic.
- Intervention (Experimental): The intervention group will receive standard of care in addition to the opportunity to access a website with engaging information about the Michigan BioTrust and a 4-minute video. Materials will be provided in English, Spanish, or Arabic.
  Interventions: Behavioral: Educational Website and Video

INTERVENTIONS:
Behavioral: Educational Website and Video — The website offers users the opportunity to choose to watch a 4-minute video or read relevant information about Newborn Screening and the Michigan BioTrust. If they choose to read, the website is designed to present information in an engaging manner, while providing optional voiceover. The video uses a mixture of live action shots and animation, all with voiceover. All materials are available in English, Spanish and Arabic.
  Arms: Intervention

SUMMARY:
The purpose of this study is to implement an electronic consent education process for the retention and research use of residual dried bloodspots at four hospitals in Michigan and assess the impact of the new education, both on patients and hospital staff. The research team will recruit women who have just given birth to answer surveys about the Michigan BioTrust consent process. Surveys will be collected from participants in the hospital and again four weeks later. The research team will collect survey data from patient participants at each hospital prior to hospital staff implementation of the new education process and again after staff implementation.

DETAILED DESCRIPTION:
The research team will compare a prospective observational control group enrolled during pre-implementation data collection within a hospital (n=2,990) to the implemented consent process group enrolled at the same hospital after implementation (2,990). Implementation will consist of hospital staff providing patients with access to a website with detailed written descriptions and a video about the Michigan BioTrust. The current standard of care, that will be maintained in addition to the new website, involves providing the patient with a brochure and descriptive information from hospital staff about the Michigan BioTrust.

A research staff member will approach patients and ask if they are willing to answer some surveys about the BioTrust consent process. After agreeing to answer the surveys, the researcher will provide them with a direct link to the research survey. If the participant does not have a phone or tablet with them, the research team member will provide a tablet upon which they can answer the questions on the survey.

All participating women or men will complete a survey 1) in the day following the BioTrust Consent and 2) at roughly 4 weeks later by email, text or telephone.

Hospital employees involved in the implementation will also answer surveys about potential sustainability immediately after completing training and again after several months of implementation.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 18 years)
* English, Spanish or Arabic speaking
* Just gave birth and currently a patient in the Mother & Baby Unit in the hospital

Exclusion Criteria:

* Parents of infants who are born pre-term (< 37 weeks gestation)
* Parents of infants in the Neonatal Intensive Care Unit
* Parents of infants being put up for adoption or in situations where legal guardianship is unknown at the time of birth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5980 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2027-11-15 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Consent and biobanking knowledge scores | Administered immediately after the intervention and at 4 week follow-up
  Knowledge will be measured with with 23 questions specific to the setting of NIPS testing, and including the multidimensional measure of informed choice (MMIC). Scored will range from 0 (no knowledge) to 23 (extremely high knowledge)
Decisional regret | Administered at the 4-week follow-up
  The Residual Decisional Regret measure assesses a person's feelings of regret after making a decision. Scores range from 1 to 5 with lower scores indicating better outcomes
Decisional Conflict | Administered immediately after the intervention and at 4 week follow-up
  The Decisional Conflict survey will determine participant uncertainty in the decision process. DCS score ranges from 0 (no decisional conflict) to 100 (extremely high decisional conflict)
Consenting rates | Obtained from the state 6 months after the end of data collection
  From the state the research team will obtain whole hospital consenting rates (people who make a decision, whether it's yes or no) for the 6-month time period before and after the Implementation
Biobanking rates | Obtained from the state 6 months after the end of data collection
  The research team will summarize the percentage who opt to participate in biobanking before and after implementation using state level data

CONTACTS AND LOCATIONS:
Overall Officials: Erin Rothwell, MD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - University of Utah Hospital and Clinics, Salt Lake City, Utah
  - University of Utah, Department of Obstetrics & Gynecology, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No